CLINICAL TRIAL: NCT02589678
Title: A Simulated Vaccine Efficacy Trial Using MMR and Tdap-IPV Vaccines in Healthy, HIV Negative Women at High Risk of HIV Infection in Lusaka and Ndola, Zambia.
Brief Title: Zambia SiVET MMR Tdap-IPV
Acronym: SiVET
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: International AIDS Vaccine Initiative (Network); Zambia-Emory HIV Research Project (Other)
Responsible Party: Principal Investigator, Susan Allen, Professor, Emory University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Screening
Other Study IDs: IRB00080202
Record Dates: First submitted 2015-10-27; First posted 2015-10-28 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: High Risk for HIV
Keywords: AIDS; Immunology; Public Health; Female sex workers; Single mothers
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Measles-Mumps-Rubella Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MMR/Tdap-IPV (Other): Participants receiving MMR vaccine (Measles, mumps, and rubella) at 0 months/at enrollment, followed by Tdap-IPV vaccine (Tetanus toxoid, reduced diphtheria toxoid and acellular pertussis) at 3 months.
  Interventions: Biological: Tdap - IPV Vaccine; Biological: MMR Vaccine
- Tdap-IPV/MMR (Other): Participants receiving Tdap-IPV vaccine (Tetanus toxoid, reduced diphtheria toxoid and acellular pertussis) at 0 months/at enrollment, followed by MMR vaccine (Measles, mumps, and rubella) at 3 months.
  Interventions: Biological: Tdap - IPV Vaccine; Biological: MMR Vaccine

INTERVENTIONS:
Biological: Tdap - IPV Vaccine — Tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine adsorbed, combined with inactivated poliomyelitis vaccine (0.5 ml) will be administered intramuscularly.
  Other Names: Adacel Quadra
Biological: MMR Vaccine — A live attenuated virus vaccine against measles, mumps and rubella (0.5 ml) will be administered intramuscularly.
  Other Names: TRIMOVAX

SUMMARY:
Participants will receive vaccination for measles, mumps, and rubella (MMR) and tetanus, diphtheria, pertussis, and inactivated polio (Tdap-IPV). The study schedule design is to simulate a vaccine efficacy trial to see if single women can participate in studies that mimic actual HIV vaccine studies.

DETAILED DESCRIPTION:
This study will evaluate if women at high risk for HIV infection residing in Lusaka, Zambia and Ndola, Zambia are willing to participate and can be retained in future HIV vaccine trials. 150 women will be enrolled that are either sex workers or single women that were identified at infant vaccination clinics (at risk due to a recent pregnancy indicating unprotected sexual contact outside of marriage or cohabitation). Two licensed vaccines will be administered as proxies for HIV vaccine administration. The clinic and laboratory procedures will simulate HIV vaccine trial procedures and will therefore inform recruitment and retention strategies and HIV incidence among high risk women in future HIV vaccine trials.

ELIGIBILITY:
Inclusion Criteria:

* At high risk of HIV, defined by occupation (female sex workers) or recent delivery (single mothers)
* Planning to stay in Lusaka or Ndola for at least 12 months
* Willing to undergo HIV testing, counseling and receive HIV test results Able and willing to provide adequate locator information for tracking purposes, and willing to be contacted by the study staff
* Willing and able to provide adequate locator information and willing to be contacted by phone if available or home visit by study staff.
* Willing to answer questions on HIV risk factors, and if infected, questions related to the route and timing of exposure
* Willing and able to return for follow-up visits
* Willing and able to provide informed consent
* Willing to undergo pregnancy testing and use an injectable, implant or intrauterine device (IUD) from screening until four months after the last vaccination during the study

Exclusion Criteria:

* HIV-1/2 infection
* Pregnant or intending to become pregnant during the study
* History of severe allergic reaction to any substance including eggs, gelatin, and neomycin
* Any clinically significant acute illness or chronic medical condition that is considered progressive, or in the opinion of the investigator, makes the volunteer unsuitable for participation in the study
* Immunosuppressive therapy
* Women who opt out of HIV counseling and testing services provided by the clinic
* Women who have any condition that in the opinion of the Investigator or designee, would preclude provision of informed consent, or otherwise interfere with achieving the study objectives
* Participation in another clinical trial unless approved by the Principal Investigator and the International AIDS Vaccine Initiative (IAVI)
* Recent receipt of an investigational blood product or vaccine
* Failure of assessment of understanding

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2015-08; Primary Completion 2017-05-16 (Actual); Study Completion 2017-05-16 (Actual)

PRIMARY OUTCOMES:
Number of participants retained | 12 Months from Baseline
  The number of participants who complete the study versus the number of participants enrolled will be calculated at the end of the study.
Number of participants who receive 1 Vaccine | 12 Months from Baseline
  The number of participants who receive at least 1 of the vaccines at the end of the study will be recorded by the study staff.
Number of participants who receive both vaccines | 12 Months from Baseline
  The number of participants who receive both vaccines at the end of the study will be recorded by the study staff.
Ratio of Female Sex Workers vs Single Mothers who adhere to study procedures | 12 Months from Baseline
  The number of female sex workers and single mothers who adhere to all study procedures will be recorded and the ratio calculated.
Number of protocol violations | 12 Months from Baseline
  The number of protocol violations that occur in the course of the study will be recorded.
Number of Corrective Action Plans | 12 Months from Baseline
  The total number of Corrective and Preventative Action Plans implemented in the course of the study to address protocol deviations will be recorded.
Time to Achieve Target Enrollment | 12 Months from Baseline
  The total time from the enrollment of first participant until enrollment of last participant will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Allen, MD, Principal Investigator — Emory University
Locations (2):
- Zambia (2):
  - Zambia Emory HIV Research Project, Lusaka
  - Zambia Emory HIV Research Project, Ndola